CLINICAL TRIAL: NCT05767970
Title: Stress Toolbox for Healthcare Providers in Mexico
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Templeton World Charity Foundation, Inc (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023-0090; Center for Healthy Minds (Other: UW Madison); L&S/PSYCHOLOGY/PSYCHOLOGY (Other: UW Madison)
Record Dates: First submitted 2023-02-28; First posted 2023-03-14 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Distress, Emotional; Burnout, Professional; Inflammation; Emotion Regulation
Keywords: Well-being
MeSH Terms: conditions — Burnout, Professional; Inflammation; Emotional Regulation | interventions — Health Personnel

STUDY DESIGN:
Intervention Model Description: Random permuted block parallel assignment
Who Masked: Investigator, Outcomes Assessor
Masking Description: Assessments will be collected online or through professional data collection service (for dried blood spots and patient satisfaction reports) that will be blind to condition assignment. The investigators responsible for data analysis will be blind to condition assignment until after primary analyses are complete.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Integrated Stress Toolbox for Healthcare Providers (ISTH) (Experimental): A 12-week synchronous and app-based well-being training that involves weekly 2-hour sessions for weeks 1-8 and at week 12, along with 12-weeks of app-based content delivered through a special version of the Healthy Minds Program app.
  Interventions: Behavioral: Integrated Stress Toolbox for Healthcare Providers (ISTH)
- Wait-list control (No Intervention): The wait-list control group will continue with business as usual and receive the ISTH after the last data collection point.

INTERVENTIONS:
Behavioral: Integrated Stress Toolbox for Healthcare Providers (ISTH) — The ISTH is a 12-week meditation-based well-being training. In weeks 1-8, participants engage in weekly 2-hour class sessions that are recorded and posted on a private Youtube channel for one week. There is a final two-hour session at week 12. In-class learning is augmented and extended through content in a special version of the Healthy Minds Program smartphone app that participants are asked to use on a daily basis throughout the intervention.
  Arms: Integrated Stress Toolbox for Healthcare Providers (ISTH)

SUMMARY:
The goal of this randomized wait-list clinical trial is to test in patient facing Mexican healthcare providers the efficacy of the Integrated Toolbox for Healthcare Providers (ISTH) on psychological functioning, well-being, occupational performance, and peripheral inflammation.

The main questions this study aims to answer are:

* Does assignment to the ISTH predict reduced psychological distress and increased well-being?
* Does assignment to the ISTH predict improved occupational outcomes and social-emotional competencies?

Participants will be randomly assigned to either the ISTH, a 12-week synchronous and app-based well-being training or to a wait-list control condition and complete assessments 8 times over the nine-month study period.

Researchers will compare the ISTH and the wait-list control group across time to evaluate ISTH impacts.

DETAILED DESCRIPTION:
Using the random permuted block method, healthcare providers from up to six Mexican states in three tiers of healthcare facilities (low, middle, and high resource) will be randomly assigned to either the 12-week ISTH intervention or wait-list control.

The ISTH consists of eight, two-hour synchronous sessions (via ZOOM) that are recorded and available to participants on a private Youtube channel for one week. Class learning is reinforced through content provided on a special version of the Healthy Mind Program app designed for this study. Weeks 8-12 of the intervention are app only, with a final two-hour synchronous session at week 12. All study content (i.e., intervention, assessments) are in Spanish.

All participants will be asked to complete a baseline assessment battery, shorter assessments after weeks 1, 3, 5, and 8, and a battery of assessments after week 12 (post-intervention), after week 24 (three-month follow-up), and after week 36 (six-month follow-up).

Researchers will randomly sample from participants opting into the dried blood spot substudy 510 participants (255 per condition) for dried blood spot collection at baseline, after week 12, and after week 24. Researchers will randomly sample from participants opting into the patient satisfaction substudy patient satisfaction reports from 4-10 of their patients at baseline, after week 12 (post-intervention) and after week 24 (three-month follow-up). Researchers will prioritize that selected participants who opted into both substudies are enrolled in the substudies.

Healthcare systems/clinics within: Nuevo León, Coahuila, Oaxaca, Querétaro, Campeche, Jalisco, and Sonora may participate.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old
* Employee in a participating healthcare system in a participating Mexican State

Exclusion Criteria:

* <18 years old
* Not in a participant healthcare system in a participating state
* Does not work in a qualifying healthcare provider role
* Does not have regular access to reliable internet and/or a smartphone capable of downloading the Healthy Minds Program app

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2315 (Actual)
Dates: Start 2023-04-04 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2025-09-29 (Actual)

PRIMARY OUTCOMES:
Change From Baseline on Psychological distress | baseline, after weeks 1, 3, 5, 8 ,12 (post intervention), 24 (3 months post-intervention), and 36 (six-months post-intervention)
  Z-scored aggregate of Patient-Reported Outcomes Measurement Information System (PROMIS) Depression (a) and Anxiety (b) Scales, and the NIH Toolbox Perceived Stress v2.0 (c). A & B: 8 item self-report scales. C: 10-item self-report. Higher scores indicate greater symptoms of psychological distress.
Change from baseline in well-being | baseline, after weeks 1, 3, 5, 8 ,12 (post intervention), 24 (3 months post-intervention), and 36 (six-months post-intervention)
  The World Health Organization Five Well-Being Index (WHO-5) is a short self-reported measure of current mental well-being (time frame the previous two weeks). The scale score range is 0 (lowest possible well-being) to 25 (highest possible well-being.

SECONDARY OUTCOMES:
Change From Baseline on the Five Facet Mindfulness Questionnaire Act With Awareness subscale | baseline, after weeks 1, 3, 8, and 12 (post intervention)
  A measure of acting with mindful awareness. Total possible scores range from 8-40, with higher scores indicating greater levels of the facet of mindfulness. This construct is specified as a mechanism of change.
Change From Baseline on the Five Facet Mindfulness Questionnaire Non-react to Inner Experience subscale | baseline, after weeks 3, 5, 8, and 12 (post intervention)
  A measure of not reacting to experience. Total possible scores range from 8-40, with higher scores indicating greater levels of the facet of mindfulness. This construct is specified as a mechanism of change.
Change from baseline on Healthy Minds Index subscales (awareness, connection, insight, and purpose) | baseline, after weeks 1, 3, 5, 8, and 12 (post intervention)
  The HM Index is a 17-item questionnaire assessing qualities trained in the HMP app (awareness, connection, insight, purpose). It is scored on a 0- to 4-point Likert scale where 0 = a low amount (e.g., never, not at all, none of the time) and 4 = a higher amount (e.g., always, to the highest degree, all of the time) of a particular quality. Total scores for the four subscales range as follows: Awareness (0 to 16), Connection (0 to 24), Insight (0 to 12), Purpose (0 to 16) where higher scores indicate more of each quality.
  Insight is specified as a mechanism of change.
Change from baseline on the Interpersonal Reactivity Index empathic concern subscale | baseline, after weeks 5, 8, and 12 (post intervention)
  A 7-item self report that measures empathic concern (i.e., compassion/care for others). It is scored on a 1-5 scale with higher scores representing greater empathic concern (score range 7 - 35).
Change from baseline on the Cognitive Emotion Regulation Questionnaire positive reappraisal subscale | baseline, after weeks 3, 5, 8, and 12 (post intervention)
  A 4-item self-report of positive reappraisal. Items are scored on a 1-5 scale (score ranges 4-20) with higher scores representing greater positive cognitive reappraisal of difficult situations. The measure is specified as a mechanism of change.
Change from baseline on the Gratitude Questionnaire-6 | baseline, after weeks 5, 8, and 12 (post intervention)
  A 6-item self-report designed to test individual differences in one's propensity to experience gratitude in daily life. Items are scored on a 1 - 7 scale, with greater scores reflecting higher levels of gratitude (score range 7 - 42).
Change from basline on the Meaning in Life Questionnaire presence subscale | baseline, after weeks 1, 8 and 12 (post intervention)
  A 5-item self report scored on a 1-7 scale, with greater score representing higher levels of meaning in life day-to-day (score ranges (5 - 35).
  This construct is specified as a mechanism.
Change from baseline on the Maslach Burnout Inventory emotional exhaustion and personal accomplishment subscales | Baseline, after weeks 8, 12 (post-intervention), 24 (three-month follow-up), and 36 (six-month follow-up)
  Burn-out is a syndrome conceptualized as resulting from chronic workplace stress that has not been successfully managed. Participants will use a 7-point frequency scale (ranging from 0-never to 6-daily) to indicate the extent to which they experienced each item (e.g., "I feel emotionally drained from my work."). Higher scores indicate higher degrees of burnout.
Change from baseline on the Multidimensional Assessment of Interoceptive Awareness (MAIA) self-regulation subscale | Baseline, after weeks 1, 3, 8, and 12 (post-intervention).
  A 4-item self-report that assess one's ability to find a sense of calm amidst feelings of overwhelm and stress. Items are scored on a 0-5 scale with higher scores representing higher levels of self-regulation (score ranges 0 - 20).
Change from baseline on the Compassionate Engagement and Action Scale Compassion for others subscale | Baseline and afters weeks 8 and 12 (post-intervention).
  A 13-item self-report that assesses compassion for others on two dimensions, engagement and action. Scores range from 13 to 130 with higher scores representing greater levels of compassion
Change from baseline on the Global Assessments of Character Strengths 24 | Baseline, after weeks 12 (post-intervention) and 36 (six-month follow-up)
  A 24 item self-report on 24 dimensions of character strengths scored on 1 - 7 scale.

OTHER OUTCOMES:
Change from baseline on peripheral inflammation assessed via dried blood spots (CRP, IL-6, IL-10, TNFalpha) | Baseline, after week 12 (post-intervention), and after week 24 (three-month follow-up)
  A four-plex of pro-inflammatory cytokines assayed via dried blood spot analytes collected in a subsample (n=525) of participants.
  Peripheral inflammation is specified as an outcome and mechanism of change.
Change from baseline on patient reports of satisfaction | Baseline and after weeks 12 (post-intervention) and 24 (three-month follow-up)
  An approximately 30 item questionnaire that a contracted agency with administer to between 4-10 patients of the subsample of participants that are enrolled in this substudy (n=525). Questions ask about overall satisfaction and levels of different provider (i.e., participant) qualities such as patience and empathy, amount of time the provider spent with the patient, quality of provider explanations, and the thoroughness of the provider's inquiry into the patients concerns.
Change from prior year to year after intervention on absenteeism. | Absenteeism year after week 24 assessment.
  Absenteeism records
Likelihood of same employment year after study | Employment year after week 24 assessment.
  Year of study and year after study employment records to test career attrition/persistence.

CONTACTS AND LOCATIONS:
Overall Officials: Leandro Chernicoff, MS, Study Director — AtentaMente
Locations (7):
- Mexico (7):
  - Campeche State, All, Campeche
  - Coahuila State, All, Coahuila
  - Jalisco State, All, Jalisco
  - Nuevo Leon State, All, Nuevo León
  - Querétaro State, All, Querétaro
  - Sonora State, All, Sonora
  - Oaxaca State, Oaxaca City

IPD SHARING:
Plan to Share IPD: Yes
Prespecified hypotheses and analyses plans will be preregistered on osf.io prior to recruitment. De-identified study data will be posted on osf.io after publication of trial analyses. Code used in all publications will be available by request.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: After publication of primary outcomes paper
Access Criteria: Data will be posted on a public repository (osf.io; e.g., to replicate published analyses) but use of the data in future publications will be at the discretion of the research team.

REFERENCES:
- [Background] Pilkonis PA, Choi SW, Reise SP, Stover AM, Riley WT, Cella D; PROMIS Cooperative Group. Item banks for measuring emotional distress from the Patient-Reported Outcomes Measurement Information System (PROMIS(R)): depression, anxiety, and anger. Assessment. 2011 Sep;18(3):263-83. doi: 10.1177/1073191111411667. Epub 2011 Jun 21. PMID 21697139
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Bech, P. (2004). Measuring the dimension of psychological general well-being by the WHO-5. Quality of Life Newsletter, 15-16.
- [Background] Maslach, C., Jackson, S. E., & Leiter, M. P. (1996). Maslach burnout inventory manual. Mountain View, CA: CPP. Inc., and Davies-Black.
- [Background] Baer RA, Smith GT, Lykins E, Button D, Krietemeyer J, Sauer S, Walsh E, Duggan D, Williams JM. Construct validity of the five facet mindfulness questionnaire in meditating and nonmeditating samples. Assessment. 2008 Sep;15(3):329-42. doi: 10.1177/1073191107313003. Epub 2008 Feb 29. PMID 18310597
- [Background] Davis, M. H. (1980). Interpersonal reactivity index.
- [Background] Garnefski, N., & Kraaij, V. (2007). The cognitive emotion regulation questionnaire. European journal of psychological assessment, 23(3), 141-149.
- [Background] Mccullough ME, Emmons RA, Tsang JA. The grateful disposition: a conceptual and empirical topography. J Pers Soc Psychol. 2002 Jan;82(1):112-27. doi: 10.1037//0022-3514.82.1.112. PMID 11811629
- [Background] Steger, M. F., Frazier, P., Oishi, S., & Kaler, M. (2006). The meaning in life questionnaire: assessing the presence of and search for meaning in life. Journal of counseling psychology, 53(1), 80.
- [Background] Mehling WE, Price C, Daubenmier JJ, Acree M, Bartmess E, Stewart A. The Multidimensional Assessment of Interoceptive Awareness (MAIA). PLoS One. 2012;7(11):e48230. doi: 10.1371/journal.pone.0048230. Epub 2012 Nov 1. PMID 23133619
- [Background] Gilbert, P., Catarino, F., Duarte, C., Matos, M., Kolts, R., Stubbs, J., ... & Basran, J. (2017). The development of compassionate engagement and action scales for self and others. Journal of Compassionate Health Care, 4, 1-24.
- [Derived] Hirshberg MJ, Davidson RJ, Velarde Arrisueno LB, Olvera Puentes JM, Bardalez XM, Gonzalez BS, Goldberg SB, Chernicoff LI; HCP-Well Study Group. Digital Well-Being Training With Health Care Professionals: A Randomized Clinical Trial. JAMA Intern Med. 2025 Aug 18;185(10):1248-56. doi: 10.1001/jamainternmed.2025.3888. Online ahead of print. PMID 40824577